CLINICAL TRIAL: NCT04986176
Title: HC-1119 Adjuvant Treatment for Hospitalized COVID-19 Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Applied Biology, Inc. (Industry)
Collaborators: Hinova Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HC-1119-DRUG-SARS-001
Record Dates: First submitted 2021-07-28; First posted 2021-08-02 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2021-07

CONDITIONS: COVID-19 Respiratory Infection
MeSH Terms: interventions — enzalutamide

STUDY DESIGN:
Intervention Model Description: Prospective, superiority, interventional, placebo-controlled, double-blinded, randomized, parallel-assignment study
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HC-1119 + Usual Care (Experimental): 4 (40mg) soft gel capsule, 160 mg total
  Interventions: Drug: HC-1119
- Placebo + Usual Care (Placebo Comparator): 4 soft gel capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HC-1119 — oral
  Arms: HC-1119 + Usual Care
Drug: Placebo — oral
  Arms: Placebo + Usual Care

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of HC-1119 as an adjuvant treatment for hospitalized COVID-19 male and female patients.

DETAILED DESCRIPTION:
This study is designed as a prospective, superiority, interventionist, placebo-controlled, double-blinded, randomized parallel assignment study. The study evaluates the efficacy and safety of HC- 1119.

Participants will be screened for eligibility; the assessment should be completed prior to any randomization to avoid screening failures to a maximum extent. Eligible participants (men and women) will be randomized 1:1 between arms (HC-1119 and placebo). HC-1119 and placebo will be administered orally.

The dosing regimen is 160 mg daily for 14 consecutive days. All patients will receive in parallel the standard treatment for COVID -19, according to the institution's protocol.

An electronic program will be used to manage randomization and drug shipment. The whole process will be handled in a manner that is blinded for the treatment received to all involved study personnel. The study follow up period will be 28 days after the first treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to the hospital with symptoms of COVID-19.
2. Male and females age ≥18 years old.
3. Confirmed positive SARS-CoV-2, through existing RT-PCR test within 7 days prior to randomization.
4. Patients with clinical status categorized of scores 4, 5, or 6 on the COVID-19 Ordinal Scale:

   * 4) Hospitalized, not requiring supplemental oxygen - requiring ongoing medical care (COVID - 19 related or otherwise);
   * 5) Hospitalized, requiring supplemental oxygen;
   * 6) Hospitalized, on non-invasive ventilation or high flow oxygen devices;
5. Participant able to swallow 4 capsules sequentially of the medication under investigation/ placebo
6. Coagulation: INR ≤ 1.5 ×ULN, and APTT ≤ 1.5×ULN
7. Women of child-bearing potential must have negative results of plasma pregnancy test (serum HCG).
8. Participant (or legally authorized representative) gives written informed consent prior to performing any study procedures.
9. Participant (or legally authorized representative) agree that participant will not participate in another COVID-19 trial while participating in this study.

Exclusion Criteria:

1. Participant enrolled in another interventionist study for COVID -19 treatment.
2. Patients requiring mechanical ventilation.
3. Patients taking an anti-androgen of any type including: androgen depravation therapy, 5-alpha reductase inhibitors, etc, having last dose of treatment less than 3 months prior to screening.
4. Patients who are allergic to the investigational product or similar drugs (or any excipients).
5. Patients has malignant tumors in the past 5 years, except for completed resected basal cell and squamous cell skin cancer and completely resected carcinoma in situ of any type.
6. Patient with known serious cardiovascular disease:

   1. Heart Failure NYHA III.
   2. Heart Failure NYHA IV.
   3. Angina class III -Canadian cardiovascular Society.
   4. Angina class IV -Canadian cardiovascular Society
   5. Angina with recent onset of symptoms, whose symptoms started 30 days or less.
   6. Myocardial infarction the last 3 months.
   7. Stroke in the last 3 months.
7. Patient with a history of seizures/epilepsy.
8. Patient taking any medications (or combination of medications) that could induce seizures/epilepsy during the study period.
9. Patient with uncontrolled medical conditions despite adequate medication, that could compromise participation in the study (e.g., uncontrolled hypertension, hypothyroidism, diabetes mellitus).
10. Known diagnosis of human immunodeficiency virus (HIV), hepatitis C, active hepatitis B, treponema pallidum (testing is not mandatory).
11. Alanine Transaminase (ALT) or Aspartate Transaminase (AST) > 5 times the upper limit of normal.
12. Estimated glomerular filtration rate (eGFR) < 30 ml/min.
13. Severe kidney disease requiring dialysis.
14. Patient likely to transfer to another hospital within 28 days after hospitalization.
15. Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless using a highly effective method of contraception (detailed in the study protocol) throughout the study and for 3 months after stopping treatment with HC-1119.
16. Sexually active men who refuse to use a condom during intercourse while taking HC-1119 and for 3 months after stopping treatment.
17. Pregnant, breastfeeding, or women planning to become pregnant 3 months after treatment with HC-1119
18. Participant (or legally authorized representative) not willing or unable to provide informed consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 602 (Estimated)
Dates: Start 2022-04-15 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality risk ratio assessed by the proportion of patient deaths in both study arms. | 28 days
  The proportion of patients reaching score 8 (death) on the COVID-19 ordinal scale at any given time up to 28 days for both study arms.

SECONDARY OUTCOMES:
Recovery ratio assessed by measuring the proportion of recovered patients in both study arms. | 28 days
  Recovery will be defined as reaching scores 1 (Not hospitalized, no limitations on activities) and 2 (Not hospitalized, limitation on activities and/or requiring home oxygen) on the COVID-19 ordinal scale.
Recovery ratio assessed by measuring the proportion of recovered patients in both study arms. | 14 days
  Recovery will be defined as reaching scores 1 (Not hospitalized, no limitations on activities) and 2 (Not hospitalized, limitation on activities and/or requiring home oxygen) on the COVID-19 ordinal scale.
Post-randomization time to recover/alive hospital discharge assessed by the median days (interquartile range) of time to recover. | 28 days
  The median days (interquartile range) of time to recover will be calculated based on the number of days subjects will lead to reach scores 1 and 2 in the COVID-19 ordinal scale.
Hazard ratio for death assessed by measuring the proportion of deaths by time in both study arms. | 28 days
  The percentage of patients that reached score 8 (death) in the COVID-19 ordinal scale at any given time up to 28 days for both study arms will allow for the calculation of the hazard ratio for death.
Pharmacokinetics of HC-1119 assessed by area under the plasma concentration-time curve from time 0 to infinity (∞) (AUC0-∞) | 14 days
Pharmacokinetics of HC-1119 assessed by area under the plasma concentration-time curve from time 0 to time t of the last measurable concentration (AUC 0-t) | 14 days
Pharmacokinetics of HC-1119 assessed by peak concentration (Cmax) | 14 days
Pharmacokinetics of HC-1119 assessed by peak time (Tmax) | 14 days
Pharmacokinetics of HC-1119 assessed by elimination half-life (t 1/2) | 14 days
Efficacy of concomitant therapies assessed by sensitivity analysis of the primary, and key secondary outcomes. | 28 days
  Sensitivity analysis of the primary, and key secondary outcomes to evaluate the efficacy of concomitant therapy including off-label use of marketed medications that are intended as treatment for COVID 19 and are given to patient prior to and during the study.

IPD SHARING:
Plan to Share IPD: No